CLINICAL TRIAL: NCT04258306
Title: Randomized, Single-blind, Cross-over Pilot Study to Evaluate the Plasma Profile of Resveratrol Following an Oral Administration of Either Revifast® (Resveratrol From Polygonum Cuspidatum Extract Siebold & Zucc - Root Supported on Magnesium Hydration With a Weight Titer of Min. 30% Resveratrol) and Unsupported Pure Resveratrol
Brief Title: Pilot Study to Evaluate the Plasma Profile of Revifast
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bernard Fioretti (Other)
Responsible Party: Sponsor-Investigator, Bernard Fioretti, Associate Professor of General Phisiology, University Of Perugia
Organization: University Of Perugia (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: RVF01
Record Dates: First submitted 2020-01-31; First posted 2020-02-06 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Nutrient; Excess; Product Use Issue
Keywords: Pharmacokinetics of resveratrol. Plasma profile of a new formulation based on resveratrol
MeSH Terms: interventions — Resveratrol

STUDY DESIGN:
Intervention Model Description: The subjects will be given, on the first day, in the morning on an empty stomach, a solution of content A or B obtained by dissolving the contents of the capsule in water which will then be taken orally. Samples of 2 ml of venous blood in a tube containing EDTA will be taken from a vein in the arm using a cannula at 0 min (fasting before administration), 15 min, 30 min, 60 min, 90 min, 120 min, 180 min. WASH-OUT on the second day. On the third day, the person who had taken the solution A will take the solution B, and vice versa, with the same methods and times described above.
Who Masked: Participant
Masking Description: Single blind, the subject, but not the responsible investigator, does not know which of the two possible treatments he receives.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resveratrol (Active Comparator): 180 mg natural Resveratrol (Polygonum cuspidatum 98%) deriving from galenic preparation from the IRRE pharmacy - Istituto Riuniti based in Cannara in via Vittorio Emanuele II 23.
  Interventions: Dietary Supplement: pure resveratrol
- REVIFAST (Experimental): 180 mg of Revifast® (mixture of resveratrol from Polygonum cuspidatum extract Siebold & Zucc. Root supported on Magnesium hydroxide).
  Interventions: Dietary Supplement: Revifast

INTERVENTIONS:
Dietary Supplement: Revifast — Revifast® is based on natural resveratrol supported on Magnesium hydroxide. Revifast® particles confer an improved dissolution rate in tests that mimic the gastric environment compared to Polygonum cuspidatum resveratrol (98%).
  Arms: REVIFAST
Dietary Supplement: pure resveratrol — resveratrol extracted from Polygonum cuspidatum resveratrol (98%).
  Other Names: trans-resveratrol
  Arms: Resveratrol

SUMMARY:
The purpose of this study is to evaluate in 6 subjects aged between 18 and 60 years the peak blood (plasma profile) of two formulations, indistinguishable from each other, containing:

A) 180 mg natural Resveratrol (Polygonum cuspidatum 98%) B) 180 mg of Revifast® (resveratrol from supported on Magnesium hydroxide).

DETAILED DESCRIPTION:
The study will be randomized, controlled, single blind, cross-over, using the two granular compounds in capsules A and B, indistinguishable from each other, dissolved in aqueous solution and administered orally. either A:180 mg natural Resveratrol (Polygonum cuspidatum 98%) deriving from galenic preparation from the IRRE pharmacy - Istituto Riuniti based in Cannara in via Vittorio Emanuele II 23.

B) 180 mg of Revifast® (mixture of resveratrol from Polygonum cuspidatum extract Siebold & Zucc. Root supported on Magnesium hydroxide).

Cross-over refers to a type of clinical study in which each individual receives each of the treatments consecutively.

PHASE I: The subjects will be given, on the first day, in the morning on an empty stomach, a solution of content A or B obtained by dissolving the contents of the capsule in water which will then be taken orally. Samples of 2 ml of venous blood in a tube containing EDTA will be taken from a vein in the arm using a cannula at 0 min (fasting before administration), 15 min, 30 min, 60 min, 90 min, 120 min, 180 min .

WASH-OUT: 1 day. PHASE II: On the third day, the person who had taken the solution A will take the solution B, and vice versa, with the same methods and times described above.

The study will have a total duration of 6 weeks divided as follows:

* Pre-monitoring phase, enrollment of subjects, random assignment in two arms 1 and 2 each consisting of 3 subjects and signature of the informative consent regarding the adhesion to the study protocol (1 week);
* 1 week for taking samples and storing them for routine chemical / biochemical analyzes carried out at the Crabion S.R.L. accredited center based in Corciano in via Amilcare Ponchielli 8 (on the first day, arm 1 will start treatment with solution A; on the second day, this arm will wash-out and arm 2 will start treatment with solution A; on third day on arm 1 will start the treatment with solution B and arm 2 will wash-out; on the fourth day arm 2 will carry out the treatment with solution B; once the routine analyzes have been carried out, on the fifth day the frozen samples will be sent to the Department of chemistry, biology and biotechnology of the University of Perugia for subsequent extraroutine analyzes).
* 2 weeks for carrying out the pharmacological and metabolomic analyzes of extraroutins performed at the Department of chemistry, biology and biotechnology of the University of Perugia;
* 2 weeks for carrying out statistical tests and processing the data obtained.

ELIGIBILITY:
Inclusion Criteria:

* Subjects naive to taking resveratrol, willing and able to understand and sign an informed consent;
* Normal blood and chemical tests: blood count, lipid structure, kidney and liver function, inflammatory structure (Tnfα, reactive protein C, ESR), glycemic profile (Fasting blood glucose, HbA1C, insulinemia, Homa Index).

Exclusion Criteria:

* Chronic pathologies (chronic renal failure, chronic hepatocellular insufficiency, autoimmune diseases, chronic inflammatory bowel diseases, diabetes mellitus, end-stage neoplasms, symptomatic chronic ischemic heart disease);
* severe arterial hypertension;
* High degree hypercholesterolaemia;
* Up to two previous days' intake of red wine not exceeding 2 glasses / day for men and 1 glass / day for women;
* Up to two previous days intake of foods containing resveratrol (red grapes, blueberries, dried fruit);
* Age <18 years;
* Poor compliance;
* Taking dietary supplements containing antioxidants;
* Untreated hypothyroidism;
* Pregnant and breastfeeding women

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2017-11-20 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Evaluate the plasma concentration (micromolar concentration) of free resveratrol after administration of a tablet containing 150mg of resveratrol in either the Resv@MDH form or pure resveratrol dissolved in water. | 2 days
  Analysis of the peak plasmatic profile of resveratrol in venous blood samples at specific time intervals and after administration of a tablet dissolved in water of two different formulations based on resveratrol. Timing of blood samples: (fasting before administration), 15 min, 30 min, 60 min, 90 min, 120 min, 180 min after oral administration. Samples of blood will be analyzed for pharmacological and metabolomic analysis of resveratrol and evaluate the concentration of resveratrol (micro molar) using a mass spectrometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Deparment of Chemistry, Biology and Biotechnology, Perugia, PG, Italy

IPD SHARING:
Plan to Share IPD: No